CLINICAL TRIAL: NCT01100177
Title: An Open Label Non- Randomized Multicentric Phase II Study of Sunitinib Before and During Radiotherapy in Newly Diagnosed Biopsy-only Glioblastoma Patients
Brief Title: Study of Sunitinib Before and During Radiotherapy in Newly Diagnosed Biopsy-only Glioblastoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENOM-008
Record Dates: First submitted 2010-04-01; First posted 2010-04-08 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Glioblastoma
Keywords: Patients with non resectable Glioblastoma who have only a; biopsy as surgical treatment
MeSH Terms: conditions — Glioblastoma | interventions — Sunitinib; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib plus radiothery (Experimental): * Sunitinib at doses of 37.5mg/m2/daily in a continuous dosing during 8 weeks.
  * After evaluation of efficacy, they will receive Sunitinib 37.5 mg/d and treatment with Radiation therapy (total dose 60 Gy).
  * After radiation therapy, Sunitinib al 37.5 mg/d will be continued until progression.
  Interventions: Drug: Sunitinib; Radiation: Radiation

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 37.5mg/m2/d
Radiation: Radiation — Radiation therapy (60Gy) 2 Gy per day during 30 days

SUMMARY:
Sunitinib seems to be a promising treatment for the objective of this proposal: to evaluate the clinical activity of Sunitinib as first line therapy in patients who have measurable disease and to evaluate the safety of Sunitinib with radiation therapy.

DETAILED DESCRIPTION:
Sunitinib (SU 11248) is a small molecule with good oral bioavailability that inhibits multiple receptor tyrosine kinases (RTKs) expressed on diverse tumour cells: VEGFR, PDGFR, KIT, FLT3 and endothelium, pericytes, and stroma VEGFR, PDGFR. It has the potential to inhibit directly the growth of multiple tumour types by the inhibition of multiple targets and to act negatively on antiangiogenesis.

Glioblastoma (GB) is the most frequent brain tumour. Standard treatment after surgical resection is radiation therapy with Temozolomide. But patients who can afford only a biopsy of their lesion due to the location in eloquent areas of their tumour or multifocality, don't get benefit from such treatment and their median survival is in the best case of only 9 months. These patients constitute 30% of Glioblastomas. Clinical trials in this setting are required as patients should be treated immediately after the biopsy to prevent neurological deterioration.

These patients are ideal to test new promising therapies. Their survival is similar to recurrent patients. The evaluation of response is easier as it's possible to avoid the confounding post-surgical changes that interfere with the evaluation of treatment efficacy in terms of tumour size reduction.. Furthermore, neo adjuvant treatment before radiotherapy has shown not to worsen their survival.

Glioblastoma is a tumour rich in molecular abnormalities. PDGFRs are important in growth signalling pathways and neoangiogenesis of gliomas. PDGF ligands and PDGFR-alfa are expressed in most human gliomas, while PDGFR-beta is expressed in glioma cells and tumor endothelial cells, PDFGR-α is expressed in most human gliomas. Imatinib mesylate exhibited antiglioma activity in preclinical studies, sensitizes glioma cells to radiation injury, and combined with hydroxyurea has shown promising results in the recurrent setting.

Moreover gliomas are among the most angiogenic cancers. VEGF/VEGFR-2 is the most prominent angiogenic signalling pathway. Its inhibition either by a neutralizing anti-VEGF antibody, anti-sense VEGF constructs, expression of a dominant-negative mutant form of VEGFR-2 (a specific small molecule inhibitor of the VEGFR-2 tyrosine kinase) or neutralizing anti-VEGFR-2 antibody has resulted in suppression of experimental malignant glioma growth. VEGF has been the focus in the development of glioma-targeted therapies. Recently Bevacizumab has shown to be active in phase II studies.

For these reasons, Sunitinib seems to be a promising treatment fo The objective of this proposal is to evaluate the clinical activity of Sunitinib as first line therapy in patients who have measurable disease and to evaluate the safety of Sunitinib with radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with glioblastoma, non resectable, who have only a biopsy as surgical treatment.
2. Measurable disease and with contrast capture of 2cm
3. Stable doses of DXM during the week before the inclusion
4. Performance status 0-1-2
5. Age < 75 years
6. MMS > 25/30
7. Barthel index > 50%
8. Surgical incision must have healed before the inclusion
9. Basal MRI done 3 weeks at the most before the beginning of the treatment which has specified conditions at the protocol.
10. FEVI > 50%
11. Suitable medullar reserve (neutrophils _2000x109/L, platelets _ 100x109/L, Haemoglobin _ 10 g/dl.)
12. Not previous chemotherapy or radiation treatment.
13. Creatinin < 1,5 times the superior standard limit of the laboratory in charged of the analysis.
14. Serum Bilirubin < 1, 5/ULN, SGOT y SGPT _ 2,5 times the superior standard limit of the laboratory in charged of the analysis. Serum alkaline phosphatases < 3/ULN.
15. Effective contraception method in patients and their couple.
16. Informed consent.

Exclusion Criteria:

1. Previous radiation or chemotherapy for the glioma´s treatment.
2. Less than 5 years time from any previous infiltrant neoplasia
3. Serious Cerebral haemorrhage after biopsy
4. Anticomital treatment inducting / inhibiting the CYP3A4 enzyme: fenitoin, carbamacepzin, phenobarbitone or other drugs that interact with sunitinib metabolism and that could not be replaced by another drug without interactions with Sunitinib.
5. Pregnancy or lactation.
6. Active or not controlled cardiovascular disease such as hypertension, angor instable, cardiac congestive failure IInd degree (NYHA), cardiac arrhythmia, previous myocardium heart attack, up to 1 year before the randomization
7. Currently treatment established with therapeutic doses of derivated anticoagulants of coumarin (coumarin, warfarin) or a week before the beginning of sunitinib. The administration of heparins of low molecular weight for TVP's control is allowed
8. Patient with TVP
9. HTA with higher values than 150/100 and not controllable with antihypertensive standard drugs
10. Not healed scars, sores or bone fractures
11. Hemorrhagic diathesis or coagulate illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate to Sunitinib therapy | 8 weeks after treatment
  Clinical activity in terms of clinical response (RANO criteria) after 2, 4 weeks cycles of Sunitinib treatment.

SECONDARY OUTCOMES:
Safety of Sunitinib with Radiation therapy | 14 weeks
  Percentage of patients without neurological damage after the first 14 weeks of the treatment
Assess the number of patients without neurological deterioration before radiation | 8 weeks
Evaluation of progression free survival | participants are followed until progression
  After radiation therapy, Sunitinib will be continued until progression. (Evaluation of progression free survival)
Overall survival | participants are followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Balaña, Coordiantor, Study Chair — Hospital Germans Trias i Pujol, Badalona, Spain
Locations (1):
- Grupo Español de Investigacion en Neurooncologia, Madrid, Madrid, Spain

REFERENCES:
- See also: Related Info — http://www.geino.es